CLINICAL TRIAL: NCT02253940
Title: An Open-label, Randomized, Crossover Relative BA Study of Pharmacokinetics and Safety of New SDS-containing Tablet and Capsule Formulations of BILR 355 Compared to the Current Formulation (50 mg Tablet), After Single Dose Oral Administration of BILR 355 Plus Low Dose Ritonavir in Healthy Male Volunteers
Brief Title: Pharmacokinetics and Safety of BILR 355 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1188.33
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Dosage Forms; Ritonavir

ARMS (2):
- Dose Group 1 - low dose (Experimental): Treatment sequences ABC / CAB / BCA
  Interventions: Drug: BILR 355 - Treatment A (current tablet formulation); Drug: BILR 355 - Treatment B (new tablet formulation); Drug: BILR 355 - Treatment C (new capsule formulation); Drug: Ritonavir
- Dose Group 2 - high dose (Experimental): Treatment sequences DE / ED
  Interventions: Drug: BILR 355 - Treatment D (current tablet formulation); Drug: BILR 355 - Treatment E (new capsule formulation); Drug: Ritonavir

INTERVENTIONS:
Drug: BILR 355 - Treatment A (current tablet formulation)
  Arms: Dose Group 1 - low dose
Drug: BILR 355 - Treatment B (new tablet formulation)
  Arms: Dose Group 1 - low dose
Drug: BILR 355 - Treatment C (new capsule formulation)
  Arms: Dose Group 1 - low dose
Drug: BILR 355 - Treatment D (current tablet formulation)
  Arms: Dose Group 2 - high dose
Drug: BILR 355 - Treatment E (new capsule formulation)
  Arms: Dose Group 2 - high dose
Drug: Ritonavir

SUMMARY:
Study to determine the single dose, relative BA of new SDS-containing formulations of BILR 355 (150 mg and 200 mg capsules and 150 mg tablet), compared to the current SDS tablet formulation (50 mg tablet)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy HIV negative adult male volunteers
2. Age ≥18 and ≤60 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2
4. Ability to give signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local regulations

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Surgery of gastrointestinal tract (except appendectomy)
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy) which was deemed relevant to the trial as judged by the investigator
7. Intake of drugs with a long half-life (>24 hours) within at least one month prior to study drug administration and during the trial
8. Use of drugs within 10 days prior to administration or during the trial which might reasonably influence the results of the trial
9. Participation in another trial with an investigational drug within two months prior to administration or during the trial
10. Current smoker
11. Alcohol abuse (more than 60 g/day)
12. Drug abuse (positive urine test for illicit prescription or non-prescription drugs or drugs of abuse)
13. Blood donation (more than 100 mL within four weeks prior to study drug administration or during the trial)
14. Excessive physical activities (within one week prior to study drug administration or during the trial)
15. Any laboratory value outside the reference range that was of clinical relevance at screening, according to the judgment of the investigator
16. Inability to comply with dietary regimen required by the protocol
17. Infected with hepatitis B or hepatitis C viruses (defined as either being hepatitis B surface antigen, or hepatitis C antibody positive)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
AUC0-inf (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 96 hours after drug administration
Cmax (maximum measured concentration of analyte in plasma) | up to 96 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 96 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 96 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 96 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 96 hours after drug administration
Number of subjects with adverse events | up to 12 days following last drug administration
Number of subjects with abnormal changes in laboratory parameters | up to 48 hours after drug administration